CLINICAL TRIAL: NCT03079843
Title: Particulate Matter, Blood Pressure, and the Sympathetic Nervous System: Impact of Near-roadway Exposures and N-95 Facemasks
Brief Title: Particulate Matter, Blood Pressure, and the Sympathetic Nervous System
Acronym: PM-SNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Robert Brook, Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HUM00122766
Record Dates: First submitted 2017-02-10; First posted 2017-03-15 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Air Pollution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- facemask first then no face mask (Experimental): wearing of mask each day for the two hours of exposure for the first week of exposure then not wearing the mask each day for the two hours of exposure for the second week of exposure
  Interventions: Other: exposure to particulate matter with N 95 facemask; Other: exposure to particulate matter with no face mask
- no face mask followed by wearing face mask (Experimental): not wearing the mask each day for the two hours of exposure for the first week of exposure then wearing the mask each day for the two hours of exposure for the second week of exposure
  Interventions: Other: exposure to particulate matter with N 95 facemask; Other: exposure to particulate matter with no face mask

INTERVENTIONS:
Other: exposure to particulate matter with N 95 facemask — 2 hours' / day exposure to particulate matter face mask worn during exposure.
  Other Names: Dettol PROTECT+ Smart Mask
Other: exposure to particulate matter with no face mask — 2 hours'/ day exposure to particulate matter with no face mask

SUMMARY:
Healthy volunteers will be exposed to ambient air near a roadway under the conditions of with and without a facemask and their responses will be evaluated.

DETAILED DESCRIPTION:
The investigators will enroll 50 healthy nonsmoking adults (20-65 years old) into a protocol involving 2 separate 5 day long "study blocks". Each block will consist of 5 separate 2 hour-long "exposure periods" conducted 5 days in a row (Monday - Friday; start: 8 am to end: 10 am) (Table 2: Study flow chart). Investigators will enroll 2 patients to undergo the trial study blocks simultaneously (one subject starting block 1 in the active intervention by wearing the facemask and the other wearing no facemask to begin block 1). Day 1 (Monday) of each study block will occur in a non-polluted clean indoor setting (Research Exam Room, Suite A 1310; Lobby A, Dominos Farms). All subsequent exposure periods (days 2-5, Tuesday through Friday) of each study block will all take place at the same designated "exposure site", an Ann Arbor Transportation Association (AATA) parking lot area nearby several busy roadways in Ann Arbor MI. To complete the entire study, each subject will perform 2 separate study blocks. Minimal total study duration is 2 weeks (washout period = 2 days over weekend) to a maximal period of 6 weeks (wash out period = 5 weeks). During one block, subjects will wear an N-95 respirator facemask (active intervention) during all exposure periods (days 1-5, even during day 1 indoor exposures). Subjects will remove the mask at the end of the study day after all testing is completed. Active versus control intervention ordering will be performed in a randomized single-blind cross-over order. During the other block subjects will wear no facemask (control) during exposure periods. While subjects will necessarily be aware of the intervention type, the study investigators responsible for evaluating the results will be blinded to the intervention type during all data analyses (i.e., single blind trial). Throughout all exposure periods, subjects will wear ambulatory BP monitors (ABPM) and ECG Holter monitors to determine brachial BP/aortic hemodynamics measured every 10 minutes and heart rate variability (HRV) metrics measured continuously and averaged into 10 minute epochs corresponding to same time periods as the BP levels, respectively. Air pollution exposures (PM2.5, black carbon (BC), and ultrafine particle (UFP) count), ambient temperature levels, and noise intensity will be measured continuously at the near-roadway exposure site during all exposure periods (Days 2-5). All environmental exposure metrics will also be averaged into 10 minute epochs during the exposure periods corresponding to the health outcome times. Following completion of exposure periods on day 4 (Thursday), subjects will have endothelial function measured by endoPAT (RHI) immediately post-exposures at the near-roadway site, after lying supine resting 5 minutes on a portable support. Patients will wear facemask throughout RHI testing when in the active intervention block. On the final day 5 of each study block, all subjects will have blood drawn. A sub-group (n=20) of subjects (enrolled on a first-come basis) will have SNS activity measured by MSNA. After blood draws on each study visit day subjects will remove the facemasks and can thereafter carry on with their routine daily activities. However, subjects will be asked to not deviate from their usual lifestyle during each study block. Subjects will be specifically directed to not significantly change their lifestyle (e.g., diet, sleep patterns) and/or any routine activity (e.g., exercise regimen, work, commutes, travel) throughout each study block.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-65 years old. People older than 65 years are excluded as the impact of PM2.5 on their BP is not known from our prior studies (which included younger individuals) and they have age-related increases in BP and SNS activity which may alter their associations with PM2.5 exposures and thus produce too heterogeneous a population to evaluate the linkages between PM2.5 and health outcomes.
* 2. Self-reported nonsmoker (100% abstinence for at least 1 year) living in non-smoking households (no one living in the household that smokes indoors) and no known routine exposures to air pollutants by known point sources at home, travel or occupationally (e.g., fumes, dust, secondhand smoke). Smoking and other exposures may alter any effect that ambient PM2.5 has on the health outcomes.
* 3. Able to understand the informed consent, legally provide informed consent, and able to participate for the entire duration of the study.

Exclusion Criteria:

* 1. Any facial hair (beard or mustache) that does not allow for proper fitting and air tight seal of the N95 facemask during the study that would compromise the ability of the mask to prevent exposures.
* 2. Any prior cardiovascular diseases (coronary artery disease (CAD), congestive heart failure (CHF), stroke, peripheral arterial disease (PAD), aneurysms, any revascularization)*
* 3. Prior diagnosis of hypertension, diabetes, sleep apnea*
* 4. Prior diagnosis of chronic lung diseases (asthma, chronic obstructive lung disease (COPD))*
* 5. Prior diagnosis of neurological disorders (Parkinson's disease, autonomic failure, peripheral neuropathy, seizure disorder) or other conditions at discretion of investigators*
* 6. Prior diagnosis of chronic kidney disease, any type of dialysis*
* 7. Active or history of any known cancer*
* 8. History of HIV*
* 9. Being treated for any infection with antibiotics within past month*
* 10. Mental health issue(s) including anxiety disorders, mood disorders, schizophrenia, or other conditions at discretion of investigators*
* 11. Prior diagnosis of any other chronic or acute medical condition(s) at discretion of investigators that may lead to alteration of baseline SNS activity, BP, or insulin sensitivity and thereby potentially impact the association of PM2.5 with study outcomes.
* 12. Medications for high BP or that alter BP. Any medications for cholesterol (e.g., statins). Any medications that alter blood glucose (e.g., diabetes medication)*.
* 13. Any medications or over the counter pills that may alter the association between ambient PM2.5 and the health outcomes of BP, SNS activity and insulin sensitivity by discretion of investigators*. No over the counter pills taken on routine basis (>2 times per week as standing dosage) including: anti-oxidants (vitamin C, E), NSAIDS, fish oil supplements, folic acid supplements, multivitamins, or other over the counter pills, herbs, or complimentary therapies under the discretion of the investigators. These pills can be stopped for 3 months on an elective basis and then the individual can enter the study. Other medications for chronic stable conditions that are not listed in exclusion criteria and that are not likely to influence the study results can be taken or continued as long as their doses have been stable for 3 months prior to entering the study. Estrogen or birth control can be used (any type) as long as the dosing has been stable for past 3 months. Medications or over the counter drugs used on an as needed basis (such as Tylenol or aspirin) are fine as long as not routinely taken >2 times per week)* Planned major change in lifestyle including work, activity, exercise, diet, weight during course of study*
* 14. Screening visit BP ≥140/90 mm Hg (as measured by the automated office BP device- BpTru)
* 15. Screening visit arm circumference ≥17 inches (makes home BP monitoring inaccurate as the cuff of the commercially-available devices will not fit).
* 16. Screening visit pregnancy (positive urine pregnancy test in women <50 years of age) and any plan to become pregnant during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
blood pressure | one week
  increased blood pressure as a result of air pollution exposure without the mask.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Brook, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No